CLINICAL TRIAL: NCT01270607
Title: Acupuncture and Pain Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04132010-5662
Record Dates: First submitted 2010-04-14; First posted 2011-01-05 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Acupuncture Therapy

ARMS (1):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Treatment given twice per week for 4 weeks

SUMMARY:
The purpose of this study is to test the hypothesis that acupuncture will reduce Fibromyalgia pain, via alterations in the processing of pain in the central nervous system.

DETAILED DESCRIPTION:
Patients and healthy controls will be enrolled in the study for a total of 6 weeks. This includes a screening and baseline visit, 8 acupuncture treatments (2 per week for 4 weeks), and a follow-up visit and treatment 1 week after completion of the study treatment sessions. To determine the effects of acupuncture on pain, patients and healthy controls will undergo psychophysical pain testing at four points throughout the study: Baseline (appointment 1), post-treatment 1 (appointment2), post treatment 8 (appointment 9), and at the final follow-up session (1 week from last treatment - appointment 10).Participants will also fill out a brief report on pain, sleep, and functioning on a palm pilot. This is expected to take less than 2 minutes per day and will occur throughout the 6 week study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Fibromyalgia patient OR healthy control
3. No current opioid use
4. Patients: must have had Fibromyalgia for 6 months or longer

Exclusion Criteria:

1. Inflammatory disorder (lupus, rheumatoid arthritis)
2. Current untreated depression
3. Active infection
4. Healthy controls: pain disorder or major medical condition that in the discretion of the investigator interfere with the validity of the study
5. Heart disease or use of a cardiac pacemaker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pain rating to Temporal Summation and Diffuse Noxious Inhibitory Control (DNIC) as measured by a visual analogue scale | Measured at last study acupuncture session (6 weeks post enrollment)

SECONDARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire | Change from first to last study treatment session (6 weeks)
Change in Brief Pain Inventory | Change from first to last treatment session (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States